CLINICAL TRIAL: NCT05053126
Title: A Phase 4 Randomized Double-Blind Double-Dummy Placebo & Active-Controlled Single-Dose Six-Way Crossover Study Evaluating the Abuse Potential of Lyrica® Taken Orally With Oxycodone HCL in Healthy Non-Drug Dependent Recreational Opioid Users
Brief Title: Study Evaluating Abuse Potential of Lyrica® in Healthy Non-Drug Dependent Recreational Opioid Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Viatris Specialty LLC (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: A0081365
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Abuse Potential
Keywords: Lyrica; Pregabalin; Oxycodone; Opioid; Abuse liability
MeSH Terms: interventions — Pregabalin; Oxycodone

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, double-dummy, placebo- and active-controlled, 6-treatment, 6-period crossover, single-dose, Williams square design study in healthy male and/or female adult, non drug-dependent recreational opioid users.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Lyrica 300 mg (Experimental): Single Dose
  Interventions: Drug: Pregabalin 300mg
- Lyrica 450 mg (Experimental): Single Dose
  Interventions: Drug: pregabalin 450 mg
- Lyrica 300mg with Oxycodone 20 mg (Experimental): Single Dose
  Interventions: Drug: Pregabalin 300 mg with oxycodone 20 mg
- Lyrica 450 mg with Oxycodone 20 mg (Experimental): Single Dose
  Interventions: Drug: pregabalin 450 mg with oxycodone 20 mg
- Oxycodone 20 mg (Active Comparator): Single Dose
  Interventions: Drug: oxycodone 20 mg
- Placebo (Placebo Comparator): Single Dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin 300mg — Participant will receive an oral dose of pregabalin 300 mg
  Arms: Lyrica 300 mg
Drug: pregabalin 450 mg — Participant will receive an oral dose of pregabalin 450 mg
  Arms: Lyrica 450 mg
Drug: Pregabalin 300 mg with oxycodone 20 mg — Participant will receive an oral dose of pregabalin 300 mg and oxycodone 20 mg
  Arms: Lyrica 300mg with Oxycodone 20 mg
Drug: pregabalin 450 mg with oxycodone 20 mg — Participant will receive an oral dose of pregabalin 450 mg and oxycodone 20 mg
  Arms: Lyrica 450 mg with Oxycodone 20 mg
Drug: oxycodone 20 mg — Participant will receive an oral dose of oxycodone 20 mg
  Arms: Oxycodone 20 mg
Drug: Placebo — Participant will receive an oral dose of placebo
  Arms: Placebo

SUMMARY:
This is a Phase 4 clinical study in healthy non-drug dependent recreational opioid users to assess the abuse potential of Lyrica when taken alone or in combination with oxycodone.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, placebo- and active-controlled, 6-treatment, 6-period crossover, single-dose study in healthy male and/or female adult, non drug-dependent recreational opioid users. The study includes Screening, a Qualification Phase, a Treatment Phase and Follow-up. This study will randomize approximately 60 adult male and female (at least 20% female) participants (10 participants in each sequence) in the Treatment Phase to ensure at least 48 participants complete the Treatment Phase of the study. There will be 8 visits to the clinic in total and a follow-up telephone call at the end of the study. The duration of participation will be approximately 16 weeks and 7 of the visits will involve clinic stays of 4 days/3 nights.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of screening. There must be no less than 20% female participants in the Treatment Phase.
2. Male and female participants who are overtly healthy. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, vital signs, 12-lead ECG, and/or clinical laboratory tests.
3. Participants must have drug abuse experience with opioids; ie, must have used opioids for non-therapeutic purposes (ie, for psychoactive effects) on at least 10 occasions within the last year and at least once in the 8 weeks before the Screening Visit (Visit 1).
4. Participants must satisfactorily complete both the Naloxone Challenge and the Drug Discrimination.
5. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
6. Body mass index (BMI) of 17.5 to 34 kg/m2, inclusive; and a total body weight

   ≥50 kg (110 lb).
7. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD).

Exclusion Criteria:

1. Current or past diagnosis of any type of drug dependence within the past year. Diagnosis of substance and/or alcohol dependence (excluding caffeine and nicotine) will be assessed by the Investigator using the Diagnostic and Statistical Manual-4 (DSM-4) criteria performed at Screening. Current drug use will be allowed if the candidate can produce a negative urine sample and are free of any signs/symptoms of withdrawal. The candidate will be informed if they have a positive breathalyzer test.
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
3. Any condition possibly affecting drug absorption (eg, gastrectomy) excluding cholecystectomy within 1 year prior to study.
4. Abnormal baseline EtCO2 <35mm Hg or >45 mm Hg.
5. Clinical or laboratory evidence of active hepatitis A infection or a history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C and/or positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb).
6. Participants with active suicidal ideation or suicidal behavior within 5 year prior to Screening as determined through the use of the Columbia-Suicide Severity Rating Scale (C-SSRS) or active ideation identified at Screening or on Day 0.
7. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
8. Patients with: sleep apnea, myasthenia gravis and glaucoma.
9. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
10. Herbal supplements and herbal medications must be discontinued at least 28 days prior to the first dose of study medication.
11. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives (whichever is longer) preceding the first dose of investigational product used in this study.
12. Positive urine drug screen (UDS) for substances of abuse at each admission in the Qualification and Treatment Phase, excluding tetrahydrocannabinol (THC). If a participant presents with a positive UDS excluding THC at any admission or any visit, the investigator, at his/her discretion, may reschedule a repeat of UDS until the UDS is negative, excluding THC, before the participant is permitted to participate in any phase of the study.
13. Unable to abstain from using THC during the Qualification and Treatment Phase of the study.
14. Has participated in, is currently participating in, or is seeking treatment for substance-and/or alcohol-related disorders (excluding nicotine and caffeine).
15. Has a positive alcohol breathalyzer or urine test at each admission to the study center during qualification and treatment phase. Positive results may be repeated and/or participants re-scheduled at the Investigator's discretions.
16. Participants are heavy smokers or users of other types of nicotine products (>20 cigarettes equivalents per day).
17. Participants are unable to abstain from smoking for at least 2 hours before and at least 8 hours after study drug administration.
18. Screening sitting blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes rest. If BP is ≥140 mm Hg (systolic) or

    ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility. Repeated BP tests should be spaced at least 5 minutes apart.
19. Baseline (screening) 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval as determined by the Fridericia method (QTcF) >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
20. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level 1.5 × upper limit of normal (ULN); Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
21. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
22. History of sensitivity to heparin or heparin-induced thrombocytopenia.
23. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
24. History of hypersensitivity to pregabalin or oxycodone or any of the components in the formulation of the study products.
25. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Sponsor employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dik WH Ng, PhD, Study Director — Mylan Pharmaceutials
Locations (1):
- Hassman Research Institute, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were entered into a Qualification phase involving a naloxone challenge test (to exclude subjects who were opioid dependent) and a drug discrimination test (to confirm they can tell the difference between oxycodone and placebo). Only subjects who passed the tests in the Qualification phase were randomized into the Treatment phase where they received the 6 different single dose study treatments, each separated by a washout of at least 4 days, in the order specified for Sequences 1-6 below
Groups:
- Sequence 1: Period 1: Placebo; Period 2: Oxycodone HCl 20 mg; Period 3: Pregabalin 450 mg plus Oxycodone HCl 20 mg; Period 4: Pregabalin 300 mg; Period 5: Pregabalin 300 mg plus Oxycodone HCl 20 mg; Period 6: Pregabalin 450 mg
- Sequence 2: Period 1: Oxycodone HCl 20 mg; Period 2: Pregabalin 300 mg; Period 3: Placebo; Period 4: Pregabalin 450 mg; Period 5: Pregabalin 450 mg plus Oxycodone HCl 20 mg; Period 6: Pregabalin 300 mg plus Oxycodone HCl 20 mg
- Sequence 3: Period 1: Pregabalin 300 mg; Period 2: Pregabalin 450 mg; Period 3: Oxycodone HCl 20 mg; Period 4: Pregabalin 300 mg plus Oxycodone HCl 20 mg; Period 5: Placebo; Period 6: Pregabalin 450 mg plus Oxycodone HCl 20 mg
- Sequence 4: Period 1: Pregabalin 450 mg; Period 2: Pregabalin 300 mg plus Oxycodone HCl 20 mg; Period 3: Pregabalin 300 mg; Period 4: Pregabalin 450 mg plus Oxycodone HCl 20 mg; Period 5: Oxycodone HCl 20 mg; Period 6: Placebo
- Sequence 5: Period 1: Pregabalin 300 mg plus Oxycodone HCl 20 mg; Period 2: Pregabalin 450 mg plus Oxycodone HCl 20 mg; Period 3: Pregabalin 450 mg; Period 4: Placebo; Period 5: Pregabalin 300 mg; Period 6: Oxycodone HCl 20 mg
- Sequence 6: Period 1: Pregabalin 450 mg plus Oxycodone HCl 20 mg; Period 2: Placebo; Period 3: Pregabalin 300 mg plus Oxycodone HCl 20 mg; Period 4: Oxycodone HCl 20 mg; Period 5: Pregabalin 450 mg; Period 6: Pregabalin 300 mg
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 9 | 10 | 9
Not Completed | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants who were randomized to a treatment sequence in the Treatment Phase
Groups:
- Randomized Population: All participants who were randomized to a treatment sequence in the Treatment Phase.
Arm/Group | Randomized Population
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.8 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 38
  White | 19
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Bipolar Visual Analog Scale (VAS) for "Drug Liking" Maximum Effect (Emax).
Description: Drug liking assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: up to 48 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a 100 mm scale
Groups:
- Placebo: Participants received a single oral dose of placebo
- Oxycodone 20 mg: Participants received a single oral dose of oxycodone 20 mg
- Lyrica 300 mg: Participants received a single oral dose of pregabalin 300 mg
- Lyrica 450 mg: Participants received a single oral dose of pregabalin 450 mg
- Lyrica 300mg With Oxycodone 20 mg: Participants received a single oral dose of pregabalin 300 mg and oxycodone 20 mg
- Lyrica 450 mg With Oxycodone 20 mg: Participants received a single oral dose of pregabalin 450 mg and oxycodone 20 mg
Arm/Group | Placebo | Oxycodone 20 mg | Lyrica 300 mg | Lyrica 450 mg | Lyrica 300mg With Oxycodone 20 mg | Lyrica 450 mg With Oxycodone 20 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53 | 53
Score on a 100 mm scale | 54.30 (1.786) | 90.85 (2.493) | 72.53 (3.224) | 76.05 (3.151) | 96.11 (1.559) | 95.06 (1.885)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone 20 mg; The sensitivity and integrity of the study was validated by comparing the mean responses of oxycodone HCl, the positive control (C), to the placebo (P): H0: μC - μP ≤ δ1 versus Ha: μC - μP > δ1 where δ1 =15; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 36.83, 95% CI 1-sided [lower limit 31.65], Standard Error of Mean 3.132
Statistical Analysis 2: Comparison: Placebo vs Oxycodone 20 mg vs Lyrica 300mg With Oxycodone 20 mg; The primary analysis evaluated whether pregabalin plus oxycodone HCl (T) produced mean responses that showed abuse potential that was no higher than oxycodone HCl (C). The margin for showing no significant difference was defined as 20% of the difference between oxycodone HCl (C) and Placebo (P): H0: μT - μC ≥ 0.2(μC - μP) versus Ha: μT - μC <0.2(μC - μP); Test type: Non-Inferiority — Non-inferiority margin = 0; p = 0.2469, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 1-sided [upper limit 3.4], Standard Error of Mean 3.49
Statistical Analysis 3: Comparison: Placebo vs Oxycodone 20 mg vs Lyrica 450 mg With Oxycodone 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority margin = 0; p = 0.1756, Mixed Models Analysis; Mean Difference (Final Values) = -3.3, 95% CI 1-sided [upper limit 2.5], Standard Error of Mean 3.48
Statistical Analysis 4: Comparison: Oxycodone 20 mg vs Lyrica 300 mg; The null and alternative hypotheses for evaluating whether pregabalin (L) produced mean responses that show less abuse potential than oxycodone HCl (C) were: H0: μC - μL ≤ 0.2 (μC - 50) versus Ha: μC - μL > 0.2 (μC - 50); Test type: Non-Inferiority — Non-inferiority margin = 10; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 1-sided [upper limit 4.3], Standard Error of Mean 2.84
Statistical Analysis 5: Comparison: Oxycodone 20 mg vs Lyrica 450 mg; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority — Non-inferiority margin = 10; p = 0.0099, Mixed Models Analysis; Mean Difference (Final Values) = 3.3, 95% CI 1-sided [upper limit 8.0], Standard Error of Mean 2.84
Statistical Analysis 6: Comparison: Placebo vs Lyrica 300 mg; The null and alternative hypotheses for evaluating whether pregabalin (L) produced mean responses that show abuse potential similar to placebo(P) were: H0: μL - μp ≥ δ2 versus Ha: μL - μp < δ2 where δ2 = 11; Test type: Non-Inferiority — Non-inferiority margin = 11; p = 0.9888, Mixed Models Analysis; Mean Difference (Final Values) = 18.2, 95% CI 1-sided [upper limit 23.4], Standard Error of Mean 3.13
Statistical Analysis 7: Comparison: Placebo vs Lyrica 450 mg; [analysis description as in outcome 1, analysis 6]; Test type: Non-Inferiority — Non-inferiority margin = 11; p = 0.9997, Mixed Models Analysis; Mean Difference (Final Values) = 22.0, 95% CI 1-sided [upper limit 27.1], Standard Error of Mean 3.13

2. Secondary Outcome: Unipolar VAS for "High" - Maximum Effect (Emax)
Description: Maximum effect on the 100 mm visual analog scale for the question "I am feeling high" where 0 = "not at all" and 100 = "extremely"
Time Frame: up to 48 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo | Oxycodone 20 mg | Lyrica 300 mg | Lyrica 450 mg | Lyrica 300mg With Oxycodone 20 mg | Lyrica 450 mg With Oxycodone 20 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53 | 53
Score on a 100 mm scale | 10.83 (4.020) | 85.83 (4.333) | 55.83 (6.180) | 60.43 (5.801) | 91.36 (3.237) | 92.23 (3.264)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 75.60, 90% CI 2-sided [65.79 to 85.42], Standard Error of Mean 5.948
Statistical Analysis 2: Comparison: Placebo vs Lyrica 300 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 44.84, 90% CI 2-sided [35.03 to 54.65], Standard Error of Mean 5.942
Statistical Analysis 3: Comparison: Placebo vs Lyrica 450 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 49.93, 90% CI 2-sided [40.12 to 59.75], Standard Error of Mean 5.945
Statistical Analysis 4: Comparison: Placebo vs Lyrica 300mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 80.80, 90% CI 2-sided [70.99 to 90.61], Standard Error of Mean 5.942
Statistical Analysis 5: Comparison: Placebo vs Lyrica 450 mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 81.91, 90% CI 2-sided [72.09 to 91.73], Standard Error of Mean 5.948
Statistical Analysis 6: Comparison: Oxycodone 20 mg vs Lyrica 300 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -30.8, 90% CI 2-sided [-40.6 to -20.9], Standard Error of Mean 5.948
Statistical Analysis 7: Comparison: Oxycodone 20 mg vs Lyrica 450 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -25.7, 90% CI 2-sided [-35.5 to -15.9], Standard Error of Mean 5.942
Statistical Analysis 8: Comparison: Oxycodone 20 mg vs Lyrica 300mg With Oxycodone 20 mg; Test type: Other; p = 0.3829, Mixed Models Analysis; Mean Difference (Final Values) = 5.20, 90% CI 2-sided [-4.62 to 15.01], Standard Error of Mean 5.945
Statistical Analysis 9: Comparison: Oxycodone 20 mg vs Lyrica 450 mg With Oxycodone 20 mg; Test type: Other; p = 0.2896, Mixed Models Analysis; Mean Difference (Final Values) = 6.31, 90% CI 2-sided [-3.50 to 16.11], Standard Error of Mean 5.942

3. Secondary Outcome: Bipolar VAS for "Take Drug Again"
Description: 100 mm visual analog scale at 24, 36, and 48 hours post-dose for the question "I would take this drug again" where 0 = "definitely not", 50 = "neutral", and 100 = "definitely so". The data from the 24, 36, and 48 hours postdose measurements were combined into a single overall model-adjusted value for 24 to 48 hours post-treatment timeframe by estimation from a mixed model with treatment, period, treatment sequence, time, and treatment*time as fixed effects, subject nested within sequence as a random effect. The compound symmetric covariance matrix was employed. Data from all time points were included
Time Frame: Up to 48 hours after treatment (assessments were made at the following timepoints after each treatment for this outcome measure: 24, 36, and 48 hours)
Population: Modified completer population
Measure: Least Squares Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo | Oxycodone 20 mg | Lyrica 300 mg | Lyrica 450 mg | Lyrica 300mg With Oxycodone 20 mg | Lyrica 450 mg With Oxycodone 20 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53 | 53
Score on a 100 mm scale | 53.58 (2.664) | 77.05 (2.668) | 63.98 (2.661) | 64.87 (2.669) | 77.91 (2.674) | 75.92 (2.664)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 23.47, 90% CI 2-sided [19.77 to 27.17], Standard Error of Mean 2.247
Statistical Analysis 2: Comparison: Placebo vs Lyrica 300 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 10.40, 90% CI 2-sided [6.71 to 14.09], Standard Error of Mean 2.239
Statistical Analysis 3: Comparison: Placebo vs Lyrica 450 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 11.29, 90% CI 2-sided [7.59 to 14.99], Standard Error of Mean 2.248
Statistical Analysis 4: Comparison: Placebo vs Lyrica 300mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 24.33, 90% CI 2-sided [20.62 to 28.03], Standard Error of Mean 2.251
Statistical Analysis 5: Comparison: Placebo vs Lyrica 450 mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 22.34, 90% CI 2-sided [18.65 to 26.04], Standard Error of Mean 2.245
Statistical Analysis 6: Comparison: Oxycodone 20 mg vs Lyrica 300 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -13.1, 90% CI 2-sided [-16.8 to -9.38], Standard Error of Mean 2.245
Statistical Analysis 7: Comparison: Oxycodone 20 mg vs Lyrica 450 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -12.2, 90% CI 2-sided [-15.9 to -8.47], Standard Error of Mean 2.252
Statistical Analysis 8: Comparison: Oxycodone 20 mg vs Lyrica 300mg With Oxycodone 20 mg; Test type: Other; p = 0.7051, Mixed Models Analysis; Mean Difference (Final Values) = 0.86, 90% CI 2-sided [-2.86 to 4.57], Standard Error of Mean 2.258
Statistical Analysis 9: Comparison: Oxycodone 20 mg vs Lyrica 450 mg With Oxycodone 20 mg; Test type: Other; p = 0.6160, Mixed Models Analysis; Mean Difference (Final Values) = -1.13, 90% CI 2-sided [-4.82 to 2.57], Standard Error of Mean 2.246

4. Secondary Outcome: Bipolar VAS for "Overall Drug Liking"
Description: 100 mm visual analog scale at 24, 36, and 48 hours post-dose for the question "Overall, my liking for this drug is" where 0 = "definitely not", 50 = "neutral", and 100 = "definitely so". The data from the 24, 36, and 48 hours postdose measurements were combined into a single overall model-adjusted value for 24 to 48 hours post-treatment timeframe by estimation from a mixed model with treatment, period, treatment sequence, time, and treatment*time as fixed effects, subject nested within sequence as a random effect. The compound symmetric covariance matrix was employed. Data from all time points were included
Time Frame: as for outcome 3
Population: Modified completer population
Measure: Least Squares Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo | Oxycodone 20 mg | Lyrica 300 mg | Lyrica 450 mg | Lyrica 300mg With Oxycodone 20 mg | Lyrica 450 mg With Oxycodone 20 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53 | 53
Score on a 100 mm scale | 53.74 (2.762) | 75.73 (2.766) | 60.14 (2.760) | 63.54 (2.767) | 74.86 (2.772) | 75.01 (2.762)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 21.99, 90% CI 2-sided [18.31 to 25.67], Standard Error of Mean 2.235
Statistical Analysis 2: Comparison: Placebo vs Lyrica 300 mg; Test type: Other; p = 0.0042, Mixed Models Analysis; Mean Difference (Final Values) = 6.40, 90% CI 2-sided [2.73 to 10.07], Standard Error of Mean 2.227
Statistical Analysis 3: Comparison: Placebo vs Lyrica 450 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 9.80, 90% CI 2-sided [6.12 to 13.48], Standard Error of Mean 2.236
Statistical Analysis 4: Comparison: Placebo vs Lyrica 300mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 21.12, 90% CI 2-sided [17.44 to 24.81], Standard Error of Mean 2.239
Statistical Analysis 5: Comparison: Placebo vs Lyrica 450 mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 21.27, 90% CI 2-sided [17.59 to 24.95], Standard Error of Mean 2.233
Statistical Analysis 6: Comparison: Oxycodone 20 mg vs Lyrica 300 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -15.6, 90% CI 2-sided [-19.3 to -11.9], Standard Error of Mean 2.233
Statistical Analysis 7: Comparison: Oxycodone 20 mg vs Lyrica 450 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -12.2, 90% CI 2-sided [-15.9 to -8.50], Standard Error of Mean 2.240
Statistical Analysis 8: Comparison: Oxycodone 20 mg vs Lyrica 300mg With Oxycodone 20 mg; Test type: Other; p = 0.7001, Mixed Models Analysis; Mean Difference (Final Values) = -0.87, 90% CI 2-sided [-4.56 to 2.83], Standard Error of Mean 2.246
Statistical Analysis 9: Comparison: Oxycodone 20 mg vs Lyrica 450 mg With Oxycodone 20 mg; Test type: Other; p = 0.7479, Mixed Models Analysis; Mean Difference (Final Values) = -0.72, 90% CI 2-sided [-4.40 to 2.96], Standard Error of Mean 2.233

5. Secondary Outcome: Unipolar VAS for "Any Drug Effect"
Description: 100 mm visual analog scale for the question "At this moment, I can feel any drug effects" where 0 = "not at all" and 100 = "extremely"
Time Frame: up to 48 hours after treatment
Population: Modified completer population
Measure: Least Squares Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo | Oxycodone 20 mg | Lyrica 300 mg | Lyrica 450 mg | Lyrica 300mg With Oxycodone 20 mg | Lyrica 450 mg With Oxycodone 20 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53 | 53
Score on a 100 mm scale | 2.14 (2.076) | 29.97 (2.075) | 16.68 (2.073) | 20.00 (2.075) | 36.55 (2.075) | 40.98 (2.075)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 27.82, 90% CI 2-sided [25.45 to 30.19], Standard Error of Mean 1.439
Statistical Analysis 2: Comparison: Placebo vs Lyrica 300 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 14.53, 90% CI 2-sided [12.17 to 16.89], Standard Error of Mean 1.435
Statistical Analysis 3: Comparison: Placebo vs Lyrica 450 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 17.85, 90% CI 2-sided [15.49 to 20.22], Standard Error of Mean 1.437
Statistical Analysis 4: Comparison: Placebo vs Lyrica 300mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 34.40, 90% CI 2-sided [34.40 to 36.77], Standard Error of Mean 1.438
Statistical Analysis 5: Comparison: Placebo vs Lyrica 450 mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 38.84, 90% CI 2-sided [36.47 to 41.21], Standard Error of Mean 1.440
Statistical Analysis 6: Comparison: Oxycodone 20 mg vs Lyrica 300 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -13.3, 90% CI 2-sided [-15.6 to -10.9], Standard Error of Mean 1.434
Statistical Analysis 7: Comparison: Oxycodone 20 mg vs Lyrica 450 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -9.97, 90% CI 2-sided [-12.3 to -7.61], Standard Error of Mean 1.435
Statistical Analysis 8: Comparison: Oxycodone 20 mg vs Lyrica 300mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.58, 90% CI 2-sided [4.22 to 8.94], Standard Error of Mean 1.436
Statistical Analysis 9: Comparison: Oxycodone 20 mg vs Lyrica 450 mg With Oxycodone 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 11.02, 90% CI 2-sided [8.65 to 13.38], Standard Error of Mean 1.436

ADVERSE EVENTS:
Time Frame: During the entire Treatment Phase of the study, which encompassed the time interval from admission of the subject to their first Treatment Period until 28 days after study drug dosing in their last (6th) Treatment Period, including the washout in between Treatment Periods. The total duration of the Treatment Phase for each subject was dependent on visit scheduling and whether the subject completed all 6 treatment periods, and it lasted up to approximately 13 weeks.
Description: Adverse events that occur during the washout interval between treatment visits or during the follow up after the final study drug dose will be counted under the previous treatment visit
Arm/Group | Placebo | Oxycodone 20 mg | Lyrica 300 mg | Lyrica 450 mg | Lyrica 300mg With Oxycodone 20 mg | Lyrica 450 mg With Oxycodone 20 mg
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58 | 0/58 | 0/59 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/58 | 0/59 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 2/58 | 9/58 | 1/58 | 4/59 | 4/59 | 8/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=58) | Oxycodone 20 mg (N=58) | Lyrica 300 mg (N=58) | Lyrica 450 mg (N=59) | Lyrica 300mg With Oxycodone 20 mg (N=59) | Lyrica 450 mg With Oxycodone 20 mg (N=59)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT05053126/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT05053126/SAP_001.pdf